CLINICAL TRIAL: NCT01761396
Title: Modular CBT for Reducing Anxiety and Improving Educational Outcomes
Brief Title: School-based Treatment of Anxiety Research Study (STARS)
Acronym: STARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Golda S. Ginsburg, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA00075767; R324A120405 (Other Grant/Funding Number: Institute of Educational Sciences (IES))
Record Dates: First submitted 2012-10-12; First posted 2013-01-04 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Fear; Worry; Therapy; Cognitive behavioral therapy
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT (Experimental): Cognitive behavioral therapy
  Interventions: Behavioral: CBT
- UC (Active Comparator): Usual care
  Interventions: Behavioral: UC

INTERVENTIONS:
Behavioral: CBT
  Other Names: Cognitive Behavioral therapy
  Arms: CBT
Behavioral: UC
  Other Names: Usual Care
  Arms: UC

SUMMARY:
This research is being done to compare two types of talk therapy to see which is most effective in helping school children with anxiety disorders. The investigators will compare usual care (UC) with cognitive behavioral therapy (CBT). Both therapies will be administered by the school mental health counselors to see if they help children with anxiety disorders to feel less scared or worried.

DETAILED DESCRIPTION:
This four year study involves a blocked randomized controlled trial (RCT) comparing the effectiveness of school-based CBT to usual care (UC) for approximately 375 students ages 7-17 diagnosed with an anxiety disorder. Randomization will occur at the school level and the investigators propose to conduct the study in approximately 46 schools (23 in CBT; 23 UC). Evaluations will be conducted by study staff to measure treatment progress at the end of the 12-week treatment program, at a three month follows up, and at natural termination.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 6-18 inclusively
* meet DSM-IV criteria for a primary anxiety disorder

Exclusion Criteria:

* presence of a medical or psychiatric condition contraindicating study treatment (e.g., suicidal intent)
* need more immediate or alternative treatment
* receiving psychosocial treatment for anxiety
* victim of previously undisclosed child abuse and require ongoing Department of Children and Families (DCF) supervision

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions Improvement Scale | 12 weeks post-treatment
  Improvement in Clinical Anxiety Diagnosis

SECONDARY OUTCOMES:
School Records | 12 weeks post-treatment
  Academic functioning
Teacher Report Form | 12 weeks post-treatment
  classroom behavior and performance

OTHER OUTCOMES:
Screen for Child Anxiety Related Emotional Disorders | 12 weeks post-treatment
  Additional measures of symptoms, mediators, and moderators
Children's Automatic Thoughts Scale | 12 weeks post-treatment
  Cognitive distortions related to anxiety
Woodcock-Johnson Tests of Achievement | 12 weeks post-treatment
  Academic achievement and working memory
Children's Global Assessment Scale | 12 weeks post-treatment
  Global Functioning
Brief Symptom Inventory | 12 weeks post-treatment
  Parental psychopathology
The TCU Organizational Readiness to Change | 12 weeks post-treatment
  Clinician's perceptions of workplace attributes

CONTACTS AND LOCATIONS:
Overall Officials: Golda S Ginsburg, Ph.D., Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will follow IES procedures for making de-identified data set available

REFERENCES:
- [Background] Ginsburg GS, Becker KD, Drazdowski TK, Tein JY. Treating Anxiety Disorders in Inner City Schools: Results from a Pilot Randomized Controlled Trial Comparing CBT and Usual Care. Child Youth Care Forum. 2012 Feb;41(1):1-19. doi: 10.1007/s10566-011-9156-4. PMID 22701295